CLINICAL TRIAL: NCT00285142
Title: Assessment of the Effect of Rosiglitazone on Insulin Secretion in Healthy Volunteers
Brief Title: Effect of Rosiglitazone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 7715
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2006-01

CONDITIONS: Healthy
Keywords: rosiglitazone; insulin secretion; clinical trial; healthy; persons
MeSH Terms: interventions — Rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone

SUMMARY:
To evaluate :

* acute effects of a single dose of 8 mg rosiglitazone (therapeutic dose)
* on insulin secretion and
* insulin sensitivity in 12 healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.0 and 24.0

Exclusion Criteria:

-

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2004-06; Study Completion 2004-11

PRIMARY OUTCOMES:
insulin response and insulin sensitivity assessed by 2-hours 10 mmol/l hyperglycemic clamp, started 45 min after treatment intake

SECONDARY OUTCOMES:
insulin clearance
basal glycemia and insulinemia
tolerance

CONTACTS AND LOCATIONS:
Overall Officials: PIERRE PETIT, MD-PhD, Principal Investigator — Centre d'Investigation Clinique
Locations (1):
- Centre d'Investigation Clinique, Montpellier, France

REFERENCES:
- [Derived] Farret A, Chevassus H, Roux B, Petit P, Galtier F. Direct rosiglitazone-induced modifications in insulin secretion, action and clearance: a single-dose hyperglycaemic clamp study. Diabetologia. 2007 Jul;50(7):1384-7. doi: 10.1007/s00125-007-0682-4. Epub 2007 May 8. PMID 17486315